CLINICAL TRIAL: NCT04804436
Title: Do Homeodomain Interacting Protein Kinase 2 (HIPK2) Polymorphisms rs2058265, rs6464214, and rs7456421 Associate With Nephrolithiasis in Turkish Population?
Brief Title: Protein Kinase 2 (HIPK2) Polymorphisms on rs2058265, rs6464214, and rs7456421
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Omer Gokhan Doluoglu, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Geneticstone
Record Dates: First submitted 2021-03-14; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Kidney Stone
Keywords: KSD HIPK2 gene Polymorphism
MeSH Terms: conditions — Kidney Calculi | interventions — Genetic Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with nephrolithiasis (Experimental): The real-time PCR amplification was performed in a final volume of 20μL reaction mixture, including 10 ng of genomic DNA, 5 µL of TaqMan® Universal PCR Master Mix, and 0.5 µL of 40X TaqMan® assay. Thermal cycling conditions were as follows: initial denaturation at 94℃ for 3 min, 40 cycles of 94℃ for 15 s, and 60°C for 1 min. The Rotor-Gene Q Series Software Version Q 2.3.1 (Rotor-Gene Q Series, Ziagen) was used for allelic discrimination.
  Interventions: Genetic: Genetic analysis
- Healthy control group (Experimental): he real-time PCR amplification was performed in a final volume of 20μL reaction mixture, including 10 ng of genomic DNA, 5 µL of TaqMan® Universal PCR Master Mix, and 0.5 µL of 40X TaqMan® assay. Thermal cycling conditions were as follows: initial denaturation at 94℃ for 3 min, 40 cycles of 94℃ for 15 s, and 60°C for 1 min. The Rotor-Gene Q Series Software Version Q 2.3.1 (Rotor-Gene Q Series, Ziagen) was used for allelic discrimination.
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — he real-time PCR amplification was performed in a final volume of 20μL reaction mixture, including 10 ng of genomic DNA, 5 µL of TaqMan® Universal PCR Master Mix, and 0.5 µL of 40X TaqMan® assay. Thermal cycling conditions were as follows: initial denaturation at 94℃ for 3 min, 40 cycles of 94℃ for 15 s, and 60°C for 1 min. The Rotor-Gene Q Series Software Version Q 2.3.1 (Rotor-Gene Q Series, Ziagen) was used for allelic discrimination.

SUMMARY:
In the present study investigators aimed to investigate whether homeodomain interacting protein kinase 2 (HIPK2) polymorphism is associated with renal stone formation in Turkish population or not.

One hundred and twenty nine participants with calcium nephrolithiasis and 67 sex and age-matched healthy controls were enrolled in this study. For analysis of HIPK2 polymorphism, the real-time PCR amplification was performed in a final volume of 20μL reaction mixture, including 10 ng of genomic DNA, 5 µL of TaqMan® Universal PCR Master Mix, and 0.5 µL of 40X TaqMan® assay. The Rotor-Gene Q Series Software Version Q 2.3.1 (Rotor-Gene Q Series, Ziagen) was used for allelic discrimination. Chi square test was utilized to compare the differences of the genotype and allele frequencies between patients and controls.

DETAILED DESCRIPTION:
Kidney stone incidence depends on geographical, climatic, ethnic, dietary and genetic factors. Thus the prevalence rates for urinary stones change from 1% to 20%. 1,2 Genetic polymorphism also causes nephrolithiasis. The most known polymorphic genes are the calcium-sensing receptor (CASR), vitamin D receptor (VDR), and matrix gla protein (MGP), plasminogen activator, urokinase (PLAU). 3,4 Furthermore, the concordance rate of the stone disease in monozygotic twins is substantially higher than in dizygotic ones (32.4% vs. 17.3%) demonstrating that genetic factors play a vital role in the formation of nephrolithiasis. 5 Homeodomain interacting protein kinase 2 (HIPK2) has been shown to be a new androgen receptor regulator. HIPK2 and androgen were demonstrated to mediate kidney tubular epithelial cell injury and apoptosis.

Informations on HIPK2 polymorphism about renal stone formation are newfound and inconclusive. Therefore, in this study, authors aimed to investigate whether HIPK2 polymorphism is associated with renal stone formation in Turkish population or not.

ELIGIBILITY:
Inclusion Criteria:

Patients with nephrolithiasis

Exclusion Criteria:

* Patients had a history of chronic urinary tract infection
* renal failure
* gastrointestinal diseases
* increased levels of vitamin D
* sarcoidosis
* primary hyperoxaluria
* polycystic kidney disease, gout, renal tubular acidosis, primary and secondary hyperparathyroidism.

Ages: 38 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Single nucleotide polymorphism | One year
  Single nucleotide polymorphism incidence on rs2058265, rs6464214, and rs7456421

CONTACTS AND LOCATIONS:
Overall Officials: Cavit Ceylan, Professor, Study Director — University of Medical Sciences, Ministry of Health, Ankara City Hospital, Department of Urology, Ankara, Turkey
Locations (1):
- Omer Gokhan Doluoglu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No